CLINICAL TRIAL: NCT01764503
Title: to Evaluate the Long-term Results of Endoscopic Papillectomy (EP)
Brief Title: Endoscopic Papillectomy for Early Ampullary Tumors: Long-term Results of the First Large Multicenter Prospective Study
Status: Completed | Type: Observational
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, Gincul Rodica, MD, Société Française d'Endoscopie Digestive
Other Study IDs: 24
Record Dates: First submitted 2013-01-04; First posted 2013-01-09 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Ampullary Tumors
Keywords: ampullary tumors; endoscopic treatment

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Adenoma of the ampulla of Vater is rare but represents a large proportion of benign tumors occurring in the small intestine. The symptoms are usually non specific or due to pancreaticobiliary obstruction . The diagnosis can also be made in asymptomatic patients during an upper gastrointestinal endoscopy. Finally, the adenoma can be discovered during a screening procedure in patients with Familial Adenomatous Polyposis (FAP).

It has been demonstrated that ampullary adenomas have a malignant potential mimicking the "adenoma-adenocarcinoma" sequence already described in the colon. So, a complete removal is mandatory. The only exception is represented by subnormal ampulla with low grade dysplasia (LGD) adenoma discovered during screening follow-up of FAP patients. In these cases the situation can be stable during several years leading to simple, annual or biannual surveillance. Historically, the treatment was surgical, associated with a high mortality and morbidity rate for pancreaticoduodenectomy (PD) and a high recurrence rate for transduodenal resection (26 to 43%). Endoscopic papillectomy (EP) represents an alternative for patients with a benign or at least non-invasive ampullary tumor. Unlike thermal ablative methods by laser photoablation or argon plasma destruction, EP allows adequate histologic evaluation especially in case of en-bloc resection. This technique has been increasingly used in the last decade with very promising results. Nevertheless the long-term results have mainly been reported in retrospective monocentric series.

We intended to evaluate, in the first large multicenter prospective study, the long-term results of endoscopic papillectomy.

DETAILED DESCRIPTION:
The patients where selected after duodenoscopy, biopsies and endoscopic ultrasound (EUS). Adenoma with at least low grade dysplasia (LGD) was required for inclusion. Two other criteria were needed in asymptomatic patients with LGD : - an ampullary size > 1 cm at endoscopy in case of FAP ; - two series of positive biopsies in case of sporadic tumors. EUS staging was estimated as follows : uT1 = tumor without invasion of the muscularis propria (MP) of the duodenum; uT2 = invasion of the MP without invasion of the pancreas ; uT3 = invasion of pancreas ; uN- = no suspicious lymph nodes ; uN+ suspicious lymph nodes. Finally, intraductal pancreatic and/or common bile duct (CBD) growths were estimated. Only uT1N- tumors without intraductal growth were included. Exclusion criteria were: - previously treated ampulloma; - metastatic disease at CT-scan; - advanced tumor at duodenoscopy (ulceration or induration involving the duodenal roof of the papilla) ; - advanced tumor (> uT1 and/or N+) and/or intraductal invasion at EUS - absence of adenoma on the resected specimen. Intraductal ultrasonography (IDUS) was optional. IDUS staging was considered as follows : uTm = tumor without invasion of the duodenal submucosae; uTsm = tumor with invasion of the duodenal submucosae.

Investigators were 11 experienced endoscopists (10 centers) specialized in pancreaticobiliary diseases and selected as follows: at least 4 years of endoscopic retrograde cholangiopancreatography (ERCP) practice with at least six EP in the last 3 years. The procedure was standardized: submucosal injection of saline solution was reserved to duodenal extension around the ampulla; a standard polypectomy snare was used with endocut current; resection has to be performed in one fragment, the piece-meal technique was only accepted for lesions larger than 2 cm. The size of the lesion was estimated by comparison with the opened snare. The ampullary tumor was snared at the base and constant tension was applied to the snare loop during electrocautery until the lesion was sectioned. The endoscopist had to mention if the procedure was considered complete or not. When needed, hemostasis was performed by injection of diluted adrenalin (1:10 000) and/or hemoclips. Realization of any additional procedures (stone removal, biliary or pancreatic sphincterotomy, biliary or pancreatic stent placement…) were left to the endoscopist decision and recorded. Patients were hospitalized for at least 2 days after the procedure. During the first 24 hours, fasting and proton pomp inhibitor (PPI) (+/- antibiotics) administration were recommended. Feeding was accepted on day 2 in the absence of complications and final discharge at day 3. Complications occurring after discharge were recorded when reported by other health care provider or by the patient at the subsequent FU session. We documented the complications and graded their severity according to the Consensus Criteria. Treatment of the complications was recorded. Finally, the length of hospital stay and the morbidity rate were calculated.

Size, number of fragments, and final staging were stated. In case of duodenal submucosal invasion a complementary surgery was discussed. In case of absence of tumor on the resected specimen, an experienced pathologist (JYS) performed a second reading of initial biopsies.

A first endoscopic control was performed after 4 to 8 weeks with retrieval of the eventual stents and systematic biopsies. In case of evident persistence of tumoral tissue a complementary resection was done, if possible, with a new endoscopic control 4 weeks later. Follow-up (F-U) was performed at 6, 12, 18, 24 and 36 months, including clinical examination, duodenoscopy with biopsies and EUS +/- ERCP. Therapeutic success was concluded in case of: 1) R0 resection = absence of invasion of duodenal submucosa on the resected specimen and complete excision of the lesion (no residual tumoral tissue at the first endoscopic control with biopsies, or at the second control in case of iterative resection) 2) no recurrence during long-term F-U. Therapeutic failure was defined as: - early failure in case of duodenal submucosal invasion on the resected specimen and/or positive biopsies without possibility of complementary resection at first control (or second control in case of iterative resection); - late failure in case of positive biopsies (persistence or recurrence) during the FU.

ELIGIBILITY:
Inclusion Criteria:

* Adenoma with at least low grade dysplasia (LGD) was required for inclusion

Two other criteria were needed in asymptomatic patients with LGD :

* an ampullary size > 1 cm at endoscopy in case of Familial Adenomatous Polyposis (FAP) ;
* two series of positive biopsies in case of sporadic tumors
* uT1N0 lesion at EUS (tumor without invasion of the muscularis propria (MP) of the duodenum and no suspicious lymph nodes)
* without intraductal growth (pancreatic and/or common bile duct)

Exclusion criteria were:

* previously treated ampulloma;
* metastatic disease at CT-scan;
* advanced tumor at duodenoscopy (ulceration or induration involving the duodenal roof of the papilla);
* advanced tumor (uT2 = invasion of the MP without invasion of the pancreas ; uT3 = invasion of pancreas and/or N+ suspicious lymph nodes) and/or intraductal invasion at EUS
* absence of adenoma on the resected specimen.

Exclusion Criteria:

* adenoma not confirmed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with ampullary tumor histologically confirmed
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2003-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Long-term results of Endoscopic Papillectomy (EP) for early ampullary tumor | 3 years
  To describe the curative and recurrence rate of endoscopic papillectomy for early ampullary tumor

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Gincul, MD, Principal Investigator — Société Française d'Endoscopie Digestive; Bertrand Napoleon, MD, Study Chair — Société Française d'Endoscopie Digestive
Locations (1):
- Société Française d'Endoscopie Digrestive, Paris, France

REFERENCES:
- [Derived] Napoleon B, Gincul R, Ponchon T, Berthiller J, Escourrou J, Canard JM, Boyer J, Barthet M, Ponsot P, Laugier R, Helbert T, Coumaros D, Scoazec JY, Mion F, Saurin JC; Societe Francaise d'Endoscopie Digestive (SFED, French Society of Digestive Endoscopy). Endoscopic papillectomy for early ampullary tumors: long-term results from a large multicenter prospective study. Endoscopy. 2014 Feb;46(2):127-34. doi: 10.1055/s-0034-1364875. Epub 2014 Jan 29. PMID 24477368